CLINICAL TRIAL: NCT06768840
Title: Serum s100B in Generalized Vitiligo and Its Relation to Oral Baricitinib, Narrow Band Ultraviolet (B) Therapy
Brief Title: Vitiligo, New Treatment and Serum s100B
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Eman Ahmed Osman, resident doctor, South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EAOsman
Record Dates: First submitted 2024-12-26; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Vitiligo, Generalized
Keywords: vitiligo; jak inhibitor; baricitinib; oral mini pulse; dexamethasone; phototherapy
MeSH Terms: conditions — Vitiligo | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- baricitinib (Active Comparator): group A, vitiligo patients will receive oral baricitinib plus narrow band ultraviolet rays B phototherapy for 3 to 6 months and serum s100B will be measured before the start of the treatment and after three months of the treatment.
  Interventions: Drug: Baricitinib; Radiation: Narrow Band UVB Treatment
- control (No Intervention): healthy matched controls for them serum s100B will be measured
- oral mini pulse (Active Comparator): vitiligo patients will recieve oral mini pulse therapy plus phototherapy for three to six months ,serum s100B will be measured before and three months after start of the treatment.
  Interventions: Drug: oral mini pulse; Radiation: Narrow Band UVB Treatment

INTERVENTIONS:
Drug: Baricitinib — oral baricitinib 4mg for adults and 2mg for children 10-16 years for group A
  Arms: baricitinib
Drug: oral mini pulse — pulse dose of oral dexamethasone 2.5mg for adults for two consecutive days per week and half the dose for children
  Arms: oral mini pulse
Radiation: Narrow Band UVB Treatment — narrowband ultraviolet rays B phototherapy two sessions per week
  Arms: baricitinib; oral mini pulse

SUMMARY:
vitiligo is an autoimmune depigmenting skin disorder characterized by milky white macules or patches, with 2% worldwide prevalence. Vitiligo has unexpected course that significantly influences on patient's quality of life and self-esteem.

Multiple medications have been introduced for vitiligo treatment, in this study we work on one of systemic JAK inhibitors

DETAILED DESCRIPTION:
Vitiligo, an autoimmune depigmenting disorder has a worldwide prevalence of 0.5%-2.0%. distinguished by distinct, varying-shaped depigmented macules and patches. Vitiligo is thought to be a benign condition that mostly affects appearance, although it usually has a significant negative influence on patients' quality of life and self-esteem. It may also put them at higher risk of developing skin cancer and sunburn. 85%-90% of cases are generalized vitiligo, also known as non-segmental vitiligo (NSV), which is characterized by a symmetric body distribution. A number of factors contribute to the multifactorial pathophysiology of vitiligo, including metabolic disorders, oxidative stress, hereditary vulnerability, and autoimmune response. Of these, cell-mediated immunity plays a major role in melanocytes destruction .The interferon-gamma (IFN-γ), C-X-C motif chemokine ligands (CXCL9/10), and C-X-C motif chemokine receptor (CXCR3) signaling axis (IFN-γ-CXCL9/10-CXCR3 or ICC axis) has been identified as a critical mediator for the recruitment of autoimmune CXCR3+ CD8+ T cells. High amounts of INF-γ and tumor necrosis factor alpha (TNF-α) are produced by these cells, which encourage melanocytes (MC) detachment and apoptosis. MCs detachment is prevented by inhibiting IFN-γ signaling pathway, which is regulated by Janus kinase-signal transducer and activator of transcription (JAK-STAT). Treatment goals for vitiligo include arresting, re-pigmentation of existing lesions, and maintenance of re-pigmentation. Only generic immunosuppressants, including oral and topical corticosteroids, calcineurin inhibitors, phototherapy, and surgical procedures, are available as the current traditional therapeutics for vitiligo. One of the primary lines of treatment for generalized vitiligo is narrowband ultraviolet B (NB-UVB) phototherapy, which is always enhanced by combining it with other therapies. JAK inhibitors target the JAK/STAT signaling pathway and are now approved to treat many immune diseases. It was reported that individuals with vitiligo treated with JAK inhibitors had higher rates of re-pigmentation especially when combined with ultraviolet or sun exposure. Given IFN-γ signaling is specially mediated by JAK1 and JAK 2. Baricitinib is a small molecule, which mainly targets the JAK1 and JAK2 subtypes, is already used in dermatology to treat inflammatory dermatoses that are caused by JAK/STAT signaling.

The cytosolic calcium-binding S100 protein family has a variety of intracellular and extracellular activities. A damage-associated molecular pattern protein called S100B has been suggested as a gauge of melanocyte cytotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* active generalized vitiligo patients with body surface area involved >5% excluding hands and feet
* no systemic treatment for vitiligo for the last 3 months or topical treatment received for the last 4 weeks.

Exclusion Criteria:

* acrofacial, acral, segmental or mucosal vitiligo
* patients on another immunosuppressive agent
* patients have other skin conditions (psoriasis, SLE, alopecia areata) that would interfere with evaluations of the effect of study medication on vitiligo.
* patients who suffered from systemic diseases affecting S100B (e.g. Subarachnoid hemorrhage, Alzheimer disease and inflammatory diseases) or from other dermatological diseases affecting S100B level (e.g. malignant melanoma)
* Patients immunocompromised, uncontrolled arterial hypertension, clinically serious viral, bacterial, fungal, or parasitic infection, anemia, history of thromboembolic event, cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, lymphoproliferative disease, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness.
* Pregnancy and lactation.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
serum s100B in active generalized vitiligo | at the time of enrollment
  detection of the relation of s100B to disease activity in comparison to control group, quantitative assessment of human s100B calcium-binding protein B (pg. /ml) using the available kit
the effect of treatments on s100B levels | after three months of the start of treatment
  detection the effect of baricitinib ,oral mini-pulse and phototherapy on the serum levels of s100B by measuring the difference of s100B levels before and after three months of treatment .
clinical efficacy of oral baricitinib combined with phototherapy in stopping the progression of the disease. | from the enrollment to three to six months after the start of the treatment
  -the ability of oral baricitinib combined with phototherapy in suppression the activity of the disease in comparison to the conventional treatment (oral mini pulse combined with phototherapy) will be measured using vitiligo diseases activity score (VIDA) in which +4 means highly active and 0 is stable
baricitinib combined with phototherapy in achieving satisfactory re-pigmentation. | from the enrollment to three to six months after the start of the treatment
  the clinical efficacy of baricitinib +NB-UVB in achieving satisfactory re-pigmentation will be measured using vitiligo activity and severity index (VASI) scoring system in which more than or equal 75% represent excellent response and less than 25% is poor response

SECONDARY OUTCOMES:
clinical satisfaction of the patients | after stopping treatment
  patient satisfaction will be recorded on a four-point scale as grade 4 highly satisfied grade 1 dissatisfied
side effects of treatment | from the enrollment and monthly till the stopping of treatment
  the side effects of treatments e baricitinib, oral mini pulse and phototherapy through regular following up of the patients

CONTACTS AND LOCATIONS:
Overall Officials: EMAN A OSMAN, bachelor, Principal Investigator — Qena university hospital, Qena faculty of medicine
Locations (1):
- Qena university hospital, Qena faculty of medicine, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No